CLINICAL TRIAL: NCT02534766
Title: MISSION COPD - Modern Innovative SolutionS in Improving Outcomes iN - COPD - A Comparison of Clinical Outcomes Before and After the MISSION Clinic.
Brief Title: MISSION COPD - Modern Innovative SolutionS in Improving Outcomes iN COPD
Acronym: MISSION-COPD
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: PHT/2015/71
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients who attended the MISSION COPD clinics: COPD patients who attended the MISSION COPD clinics, identified as having uncontrolled or potentially severe COPD or unrecognised COPD from GP records by the MISSION clinical team
- Health Care Professionals: Health Care Professionals who attended the MISSION COPD clinics in a professional/ clinical capacity.

SUMMARY:
MISSION is a new and novel way of delivering highly specialised Chronic Obstructive Pulmonary Disease (COPD) care and has the potential to change the way COPD care across the UK is delivered as well as services for other long term health conditions. The MISSION model has been piloted in asthma which is the subject of an ongoing research study. This is the first model of this type in COPD and the current research study aims to evaluate the outcomes of the project. This will be done in several different ways. The study is a mixed methods evaluation of the new service comparing outcomes before and after the clinic using retrospective data analysis and prospective qualitative interview. The study will be conducted at Portsmouth Hospitals NHS Trust and will recruit patients who attend MISSION COPD clinics as well as staff who attended MISSION clinics in a professional capacity.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate in detail the clinical and health economic outcomes from the MISSION COPD project. MISSION COPD is a quality improvement project funded by the Health Foundation, Foundation with additional funding from Pfizer, to trial an innovative way of finding and assessing patients with COPD and also case finding new diagnoses of COPD.

MISSION-COPD will allow swift early specialist multi-disciplinary interventions in primary care to diagnose and treat those at greatest risk, consistent with the NHS England '5-year Forward View' calling for removal of traditional primary and secondary care barriers. MISSION COPD will target COPD patients with risk factors for exacerbations and deteriorating lung function as well potential new diagnoses of COPD.

The aim of the study is to review the MISSION clinic model outcomes as well as performing qualitative interviews with patients who attended and staff who took part in the project.

Up to 150 patients who attend the MISSION COPD clinic will be recruited along with approximately 20 health care professionals. The number of patients has been decided as the number that can be seen for the project in the MISSION COPD project time and budget.

Participants will be either:

* Patients who attend MISSION COPD clinics - identified as having uncontrolled or potentially severe COPD or unrecognised COPD from GP records by the MISSION clinical team
* Health care professionals who attend the clinic in a clinical capacity.

Retrospective quantitative analysis of the data collected during the MISSION clinics will be analysed looking for COPD phenotypes and contributing co-morbidities. The data collected at the initial visit and 3 and 6 month follow up questionnaires will be analysed looking for improvement in COPD control and quality of life following the patients' attendance at MISSION clinics.

A self completion questionnaire will be filled in after the clinic by participants in the research study to assess their views on the clinic and where they would like changes to be made. A questionnaire will also be given to health care professionals to seek their views on the clinic.

Qualitative interviews will be conducted with a sample of participants, willing to take part, to explore the experiences and acceptability of the participants and health care professionals. The interviews with health care professionals will explore their thoughts on MISSION and its strengths and weaknesses as well as any suggestions for improvement.

This research is important as it will provide evidence to support the use of the MISSION clinic model for patients with COPD. It will also give us more information on the patient with COPD and any medical conditions related to their COPD so we can adapt our service to meet their needs.

The telephone and group interviews will help us understand what we are doing right and what we are doing wrong with COPD care.

ELIGIBILITY:
Inclusion Criteria - Patients:

* Male of Female, aged 18 years or above.
* Attended the MISSION clinic as a patient.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria - Patients:

- The patient is unable or unwilling to give consent

Inclusion criteria - Health Care Professionals

* Male or Female, aged 18 or above.
* Attended the MISSION clinic as a health care professional
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria - Health Care Professionals

- The health care professional is unable or unwilling to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be patients who attend MISSION COPD clinics, identified as having uncontrolled or potentially severe COPD or unrecognised COPD from GP records by the MISSION clinical team or health care professionals who attend the clinic in a clinical capacity.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
COPD control measured by number of exacerbations treated with steroids and or antibiotics for ≥3 days | 6 months previous
  To assess whether the number COPD exacerbations (prednisolone or equivalent ≥30 mg for >3 days or antibiotics for >3 days) improves in MISSION patients in the 6 months after the clinic compared with the 6 months before.
COPD control measured by number of exacerbations treated with steroids and or antibiotics for ≥3 days | 6 months
  To assess whether the number COPD exacerbations (prednisolone or equivalent ≥30 mg for >3 days or antibiotics for >3 days) improves in MISSION patients in the 6 months after the clinic compared with the 6 months before.
Number of exacerbations of COPD that require hospital admission and treatment | 6 months previous
  Number of exacerbations of COPD that require admission to hospital for treatment to assess whether hospital admissions change in the 6 months after the MISSION clinic
Number of exacerbations of COPD that require hospital admission and treatment | 6 months
  Number of exacerbations of COPD that require admission to hospital for treatment to assess whether hospital admissions change in the 6 months after the MISSION clinic

SECONDARY OUTCOMES:
COPD Assessment Test (CAT) Score | baseline
  patients will complete the CAT questionnaire to assess COPD control
COPD Assessment Test (CAT) Score | 3 months
  patients will complete the CAT questionnaire to assess COPD control
COPD Assessment Test (CAT) Score | 6 months
  patients will complete the CAT questionnaire to assess COPD control
St George's Respiratory Questionnaire (SGRQ) | baseline
St George's Respiratory Questionnaire (SGRQ) | 3 months
St George's Respiratory Questionnaire (SGRQ) | 6 months
Number of non elective GP visits for COPD | 6 month previous
  Number of non elective GP visits for COPD in the 6 months pre MISSION
Number of non elective GP visits for COPD | 6 months
  Number of non elective GP visits for COPD in the 6 months post MISSION
Number of hospital admissions for COPD | 6 month previous
  Number of hospital admissions for COPD in the 6 months pre MISSION
Number of hospital admissions for COPD | 6 months
  Number of hospital admissions for COPD in the 6 months post MISSION
Number of Emergency Department contacts for COPD | 6 month previous
  Number of Emergency Department contacts for COPD in the 6 months pre MISSION
Number of Emergency Department contacts for COPD | 6 months
  Number of Emergency Department contacts for COPD in the 6 months post MISSION
Number of out of hour (OOH) attendances/contacts for COPD | 6 month previous
  Number of out of hour attendances (OOH) contacts for COPD in the 6 months pre MISSION
Number of out of hour (OOH) attendances/contacts for COPD | 6 months
  Number of out of hour attendances (OOH) contacts for COPD in the 6 months post MISSION
Global initiative in chronic Obstructive Lung Disease (GOLD) score | Baseline
  To assess the severity of COPD by GOLD and BTS stage in the MISSION clinics
Measurement and variation of lung function. | Baseline
Assessment of eosinophilic airways inflammation | Baseline
  Assessment of eosinophilic airways inflammation by Fractional Exhaled Nitric Oxide (FeNO) Assessment.
COPD controller medication | 6 months previous
  COPD controller medication in 6 months pre MISSION.
COPD controller medication | 6 months
  COPD controller medication in 6 months post MISSION.
Number of antibiotic courses without prednisolone for lower respiratory tract infections | 6 months previous
  Number of antibiotic courses without prednisolone for lower respiratory tract infections in 6 months pre MISSION
Number of antibiotic courses without prednisolone for lower respiratory tract infections | 6 months
  Number of antibiotic courses without prednisolone for lower respiratory tract infections in 6 months post MISSION
Short acting bronchodilator (SABA) use | 6 months previous
  Short acting bronchodilator (SABA) use measured by number of inhalers prescribed in 6 months pre MISSION.
Short acting bronchodilator (SABA) use | 6 months
  Short acting bronchodilator (SABA) use measured by number of inhalers prescribed in 6 months post MISSION.
Frequency and severity of co-morbidities | Baseline
  Frequency and severity of co morbidities including anxiety and depression, dysfunctional breathing, gastro oesophageal reflux and obstructive sleep apnoea in all patients.
Medication adherence | Baseline
  Medication adherence will be measured at baseline
Medication adherence | 3 months
  Medication adherence will be measured at 3 months
Medication adherence | 6 months
  Medication adherence will be measured at 6 months
Patient activation measure | Baseline
  Patients will complete the patient activation measure questionnaire at Baseline
Patient activation measure | 3 months
  Patients will complete the patient activation measure questionnaire at 3 months
Patient activation measure | 6 months
  Patients will complete the patient activation measure questionnaire at 6 months
Investigations performed | Baseline
  Investigations performed at the MISSION COPD clinics (e.g. sputum induction, High-Resolution Computed Tomography (HRCT) chest).
Hospital Anxiety and Depression Scale (HADS) score | Baseline
  HADS scores at baseline for patients attending the MISSION clinics
Hospital Anxiety and Depression Scale (HADS) score | 6 months
  HADS scores at 6 months for patients attending the MISSION clinics
Gastroesophageal Reflux Disease Questionnaire (GERDQ) score | baseline
  GERDQ scores at baseline for patients attending the Severe COPD Assessment Clinic (SCAC)
Gastroesophageal Reflux Disease Questionnaire (GERDQ) score | 6 months
  GERDQ scores at 6 months for patients attending the Severe COPD Assessment Clinic (SCAC)
Assessment of inhaler technique and recommendations for inhaler devices. | Baseline
Smoking cessation advice | Baseline
The frequency of non-attendance at clinic | Baseline
  The frequency of non-attendance at the MISSION clinic

CONTACTS AND LOCATIONS:
Overall Officials: Professor Anoop J Chauhan, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

REFERENCES:
- [Background] Kruis AL, Smidt N, Assendelft WJ, Gussekloo J, Boland MR, Rutten-van Molken M, Chavannes NH. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2013 Oct 10;(10):CD009437. doi: 10.1002/14651858.CD009437.pub2. PMID 24108523
- [Background] Wilkinson T, North M, Bourne SC. Reducing hospital admissions and improving the diagnosis of COPD in Southampton City: methods and results of a 12-month service improvement project. NPJ Prim Care Respir Med. 2014 Aug 21;24(0):14035. doi: 10.1038/npjpcrm.2014.35. PMID 25141877
- See also: Department of Health, 2011. An outcomes strategy for people with chronic obstructive pulmonary disease (COPD) and asthma in England — https://www.gov.uk/government/uploads/system/uploads/attachment_data/file/216139/dh_128428.pdf
- See also: Public Health England, 2014. Portsmouth Unitary Authority Health Profile 2014 — http://www.google.co.uk/url?sa=t&rct=j&q=&esrc=s&source=web&cd=1&ved=0CCEQFjAAahUKEwiMnbWLlcTHAhUL6RQKHc6ZB30&url=http%3A%2F%2Fwww.apho.org.uk%2Fresource%2Fview.aspx%3FRID%3D142418&ei=JFbcVYz7GYvSU86znugH&usg=AFQjCNFAG7d96FNAi44xlQ5uWh3eRHFJmg
- See also: Public Health England, 2015. Local Tobacco Control Proflies. — http://www.tobaccoprofiles.info/profile/tobacco-control/data